CLINICAL TRIAL: NCT03044795
Title: Phase II Study With PARP Inhibitor Veliparib (ABT-888) in Patients With Increased Risk of Homologous Recombination Deficiency to Determine the Value of an (Ex-vivo) RAD51 Assay as a Biomarker
Brief Title: Response to PARP Inhibitor Predicted by the RAD51 Assay
Acronym: REPAIR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study never started
Sponsor: University Medical Center Groningen (Other)
Collaborators: AbbVie (Industry); Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201600942
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: homologous recombination deficiency; veliparib; PARP inhibitor; biomarker
MeSH Terms: conditions — Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Patients with TNBC, platinum sensitive high grade serous ovarian cancer or BRCA-mutated (non-)breast and (non-)ovarian cancer will be included prior to the RAD51 assay and treated with veliparib irrespective of the assay result. All patients, including TNBC patients, will receive veliparib monotherapy until at least the first tumor assessment after 8 weeks of treatment.
  Interventions: Drug: Veliparib
- Part B (Experimental): Only patients with a RAD51 assay HR deficiency will be included. First there will be a pre-screening procedure followed by a tumor lesion biopsy on which the RAD51 assay will be performed. In case of a RAD51 assay indicating HR proficiency, patients will not be eligible for treatment in this study and cannot be included. Patients with a RAD51 assay indicating HR deficiency will be included. Eligible patients will be treated with veliparib monotherapy until at least the first tumor assessment after 8 weeks of treatment. In case of 0/15 patients within one patient subgroup having RAD51 tests showing HR-deficiency inclusion for this sub-group will be closed.
  Interventions: Drug: Veliparib

INTERVENTIONS:
Drug: Veliparib — Subjects in part A and part B will all start treatment with oral veliparib monotherapy twice a day. Patients will receive oral veliparib BID on days 1- 21, q3 weeks. All subjects will start with veliparib 300 mg, if the subject tolerates 300 mg BID for 2 weeks, veliparib may be increased to 400 mg BID at the investigator's discretion. Subjects will self-administer the morning dose and the evening dose of veliparib approximately 12 hours after the morning dose with or without food. ANC must be above 1.5 × 109/L in order to commence a new cycle.

SUMMARY:
In tumors with a defect in the homologous recombination (HR) pathway, double-strand break repair is partly impaired. Patients with HR deficient tumors benefit from therapies that induce DNA lesions requiring HR for repair. These therapies include platinum compounds and inhibitors of the enzyme PARP-1. At this moment, selection for PARP inhibitor treatment relies on detection of germ-line or somatic mutations in the HR pathway genes BRCA1 or BRCA2. However, not all HR deficient tumors have a BRCA gene mutation, the BRCA genes can also be silenced by promoter methylation. Moreover, the HR pathway can be defective due to mutations in other HR genes. In addition, the presence of a BRCA gene mutation does not guarantee defective HR since mutations in other genes (e.g. TP53BP1) can restore HR despite the presence of a BRCA1 mutation. Since all patients with tumors that are HR deficient may benefit from PARP inhibition, better tools are required to identify these patients. Recently, a functional ex vivo test for HR deficiency (the RAD51 assay) became available for clinical use. The RAD51 assay can identify patients with functional defects in HR-repair and may predict which cancer patients are likely to benefit from PARP inhibition. The purpose of this study is to investigate whether the RAD51 assay can select patients who will benefit from treatment with the PARP-inhibitor veliparib.

ELIGIBILITY:
Inclusion Criteria:

Part A

1. ≥ 18 years of age.
2. Histologically or cytologically confirmed malignancy that is metastatic or unresectable. Subjects must have either:

   1. Non-rapidly progressive disease. This means not requiring initiation of chemotherapy (within 8 weeks), based on clinician's evaluation.
   2. No effective standard of care options.
3. Subjects must have triple negative breast cancer (maximum 10% ER expression), platinum sensitive (≥ 6 months since last platinum containing therapy) high grade serous ovarian cancer or BRCA1/2 mutated (non-)breast and (non-)ovarian cancer.
4. The subject has had a maximum of 3 prior DNA damaging agents or cytotoxic chemotherapy treatments (prior therapies with biologic agents including, IL-2, interferon, vaccines, immunostimulating agents, immune checkpoint inhibitors and signal transduction inhibitors are allowed and do not count as a cytotoxic chemotherapy treatment line). Chemotherapy received as adjuvant therapy will not be considered as prior chemotherapy when administered at least 1 year before advanced disease has been detected.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 to 1.
6. Adequate hematologic, renal and hepatic function as follows:

   * Absolute Neutrophil Count (ANC) ≥ 1500/μL.
   * Platelet ≥ 100,000/μL.
   * Hemoglobin ≥ 5.6 mmol/L.
   * Serum creatinine ≤ 1.5 × upper normal limit of institution's normal range OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
   * Bilirubin ≤ 1.5 × the upper normal limit of institution's normal range.
   * Aspartate Aminotransferase (AST) and Alanine Transaminase (ALT ≤ 2.5 ) x the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT < 5 x the upper normal limit of institution's normal range.
   * APTT must be ≤ 1.5 × upper normal limit of institution's normal range and International Normalized Ratio (INR) < 1.5 for subjects not on anticoagulant therapy. Subjects on anticoagulant (such as Coumadin) will have PTT and INR as determined by the investigator.
   * Serum pregnancy test for women of childbearing potential, including women who have had a tubal ligation; childbearing potential is defined as not having undergone surgical sterilization, hysterectomy, and/or bilateral oophorectomy, or not being postmenopausal (≥ 12 months of amenorrhea).
7. Females of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 90 days following completion of therapy.
8. Measurable disease, as defined by standard RECIST v1.1 or GCIG guidelines using ca-125 in ovarian cancer. Previously irradiated lesions should not be counted as target lesions.
9. Metastatic or locally advanced lesion(s) of which a histological biopsy can safely be obtained according to standard clinical care procedures. Boney lesions are not acceptable as biopsy site.
10. Capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by an Independent Ethics Committee (IEC) prior to the initiation of any screening or study-specific procedures.

Part B

1. ≥ 18 years of age.
2. Histologically or cytologically confirmed malignancy that is metastatic or unresectable. Subjects must have either:

   1. Non-rapidly progressive disease. This means not requiring initiation of chemotherapy (within 8 weeks), based on clinician's evaluation.
   2. No effective standard of care options.
3. Subjects with an intermediate risk of HR deficiency: head and neck cancer, non-small cell lung cancer, ER+/Grade III breast cancer, gastro-intestinal cancer, bladder cancer, ovarian cancer (not platinum sensitive high grade serous, these are eligible for part A), prostate cancer and endometrial cancer, non-small cell lung cancer (squamous histology only) with defective HR as assessed by the (ex-vivo) RAD51 assay.
4. The subject has received up to 3 prior DNA damaging agents or cytotoxic chemotherapy treatments (prior therapies with biologic agents including, IL-2, interferon, vaccines, immunostimulating agents, immune checkpoint inhibitors and signal transduction inhibitors are allowed). Chemotherapy received as adjuvant therapy (with an interval more than 1 year) will not be considered as prior chemotherapy.
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 to 1.
6. Adequate hematologic, renal and hepatic function as follows:

   * Absolute Neutrophil Count (ANC) ≥ 1500/μL.
   * Platelet ≥ 100,000/μL.
   * Hemoglobin ≥ 5.6 mmol/L.
   * Serum creatinine ≤ 1.5 upper normal limit of institution's normal ranger OR creatinine clearance ≥ 50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
   * Bilirubin ≤ 1.5 × the upper normal limit of institution's normal range.
   * AST and ALT ≤ 2.5 × the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT < 5 × the upper normal limit of institution's normal range.
   * APTT must be ≤ 1.5 × upper normal limit of institution's normal range and International Normalized Ratio (INR) < 1.5. Subjects on anticoagulant (such as Coumadin) will have PTT and INR as determined by the investigator.
   * Serum pregnancy test for women of childbearing potential, including women who have had a tubal ligation; childbearing potential is defined as not having undergone surgical sterilization, hysterectomy, and/or bilateral oophorectomy, or not being postmenopausal (≥ 12 months of amenorrhea).
7. Females of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 90 days following completion of therapy.
8. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions.
9. Metastatic or locally advanced lesion(s) of which a histological biopsy can safely be obtained according to standard clinical care procedures.
10. Capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

Both part A and B:

1. Received any anti-cancer therapy including chemotherapy, immunotherapy, anti-hormonal therapy, radiotherapy, biologic or any investigational therapy within either 28 days, or 5 half-lives of a targeted therapy (whichever is shorter), prior to the first dose of veliparib.

   * For prostate cancer, subjects receiving bisphosphonates are eligible if the subject has been on stable doses of bisphosphonates for the 2 months prior to study initiation without Grade 2 or greater toxicities. For breast cancer patients bisphosphonates are allowed.
   * For prostate cancer, Luteinizing Hormone Releasing Hormone (LHRH) analogue agents are allowed if the subject has received LHRH analogues during the 2 months prior to study initiation.
2. Has known central nervous system (CNS) metastases, unless treated properly with stable disease (without dexamethasone or with a stable or reducing dose of dexamethason) for at least 3 months prior to study entry.
3. Patients at high risk for seizure such as uncontrolled seizure disorder or focal or generalized seizure within the last 12 months.
4. Clinically significant and uncontrolled major medical condition(s) including but not limited to:

   * Active uncontrolled infection.
   * Subject has previous or current malignancies at other sites, with the exception of:

     * Adequately treated in situ carcinoma of the cervix uteri;
     * Basal or squamous cell carcinoma of the skin;
     * Previous malignancy (e.g., localized prostate cancer) confined and surgically resected, treated with chemotherapy or radiation therapy, and is considered cured by the investigator.
   * Symptomatic congestive heart failure.
   * Unstable angina pectoris or cardiac arrhythmia.
   * Psychiatric illness/social situation that would limit compliance with study requirements.
   * QTc with Frederichs correction >470 ms.
   * Any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities.
5. Pregnant or breastfeeding female.
6. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive veliparib .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Part A: determine the value of the RAD51 assay in predicting response to veliparib | 8 weeks
  To determine the value of the RAD51 assay in predicting response to veliparib at eight weeks in patients with a high risk of HR deficiency.
Part B: determine response to veliparib at eight weeks in novel patient groups with HR deficient tumors a | 8 weeks
  To determine response to veliparib at eight weeks in novel patient groups with HR deficient tumors as assessed by the RAD51 assay.

CONTACTS AND LOCATIONS:
Overall Officials: J. A. Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: No